CLINICAL TRIAL: NCT03131440
Title: Designing With Dissemination in Mind: Optimization of a mHealth Physical Activity Intervention for Breast Cancer Survivors
Brief Title: Optimization of Remotely Delivered Physical Activity Intervention for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Siobhan M Phillips, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: K07CA196840 (NIH); K07CA196840 (NIH); R21CA219028-01A1 (NIH)
Record Dates: First submitted 2017-04-18; First posted 2017-04-27 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer Female; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Amyloid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Experimental Condition #1 (Experimental): core, support calls
  Interventions: Behavioral: Core; Behavioral: Support Calls
- Experimental Condition #2 (Experimental): core, support calls, app+
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App+
- Experimental Condition #3 (Experimental): core, support calls, buddy
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: Buddy
- Experimental Condition #4 (Experimental): core, support calls, online gym
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: Online gym
- Experimental Condition #5 (Experimental): core, support calls, app notifications
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App notifications
- Experimental Condition #6 (Experimental): core, app+
  Interventions: Behavioral: Core; Behavioral: App+
- Experimental Condition #7 (Experimental): core, app+, buddy
  Interventions: Behavioral: Core; Behavioral: App+; Behavioral: Buddy
- Experimental Condition #8 (Experimental): core, app+, online gym
  Interventions: Behavioral: Core; Behavioral: App+; Behavioral: Online gym
- Experimental Condition #9 (Experimental): core, app+, app notifications
  Interventions: Behavioral: Core; Behavioral: App+; Behavioral: App notifications
- Experimental Condition #10 (Experimental): core, buddy
  Interventions: Behavioral: Core; Behavioral: Buddy
- Experimental Condition #11 (Experimental): core, buddy, online gym
  Interventions: Behavioral: Core; Behavioral: Online gym; Behavioral: Buddy
- Experimental Condition #12 (Experimental): core, buddy, app notifications
  Interventions: Behavioral: Core; Behavioral: App notifications; Behavioral: Buddy
- Experimental Condition #13 (Experimental): core, online gym
  Interventions: Behavioral: Core; Behavioral: Online gym
- Experimental Condition #14 (Experimental): core, online gym, app notifications
  Interventions: Behavioral: Core; Behavioral: Online gym; Behavioral: App notifications
- Experimental Condition #15 (Experimental): core, app notifications
  Interventions: Behavioral: Core; Behavioral: App notifications
- Experimental Condition #16 (Experimental): core, support calls, app+, buddy
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App+; Behavioral: Buddy
- Experimental Condition #17 (Experimental): core, support calls, app+, online gym
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App+; Behavioral: Online gym
- Experimental Condition #18 (Experimental): core, support calls, app+, app notifications
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App+; Behavioral: App notifications
- Experimental Condition #19 (Experimental): core, support calls, buddy, online gym
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: Online gym; Behavioral: Buddy
- Experimental Condition #20 (Experimental): core, support calls, buddy, app notifications
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App notifications; Behavioral: Buddy
- Experimental Condition #21 (Experimental): core, support calls, online gym, app notifications
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: Online gym; Behavioral: App notifications
- Experimental Condition #22 (Experimental): core, app+, buddy, online gym
  Interventions: Behavioral: Core; Behavioral: App+; Behavioral: Online gym; Behavioral: Buddy
- Experimental Condition #23 (Experimental): core, app+, buddy, online gym, app notifications
  Interventions: Behavioral: Core; Behavioral: App+; Behavioral: Online gym; Behavioral: App notifications; Behavioral: Buddy
- Experimental Condition #24 (Experimental): core, support calls, buddy, online gym, app notifications
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: Online gym; Behavioral: App notifications; Behavioral: Buddy
- Experimental Condition #25 (Experimental): core, buddy, online gym, app notifications
  Interventions: Behavioral: Core; Behavioral: Online gym; Behavioral: App notifications; Behavioral: Buddy
- Experimental Condition #26 (Experimental): core, app+, online gym, app notifications
  Interventions: Behavioral: Core; Behavioral: App+; Behavioral: Online gym; Behavioral: App notifications
- Experimental Condition #27 (Experimental): core, support calls, app+, buddy, online gym
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App+; Behavioral: Online gym; Behavioral: Buddy
- Experimental Condition #28 (Experimental): core, support calls, app+, buddy, app notifications
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App+; Behavioral: App notifications; Behavioral: Buddy
- Experimental Condition #29 (Experimental): core, support calls, app+, online gym, app notifications
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App+; Behavioral: Online gym; Behavioral: App notifications
- Experimental Condition #30 (Experimental): core
  Interventions: Behavioral: Core
- Experimental Condition #31 (Experimental): core, app+, buddy, app notifications
  Interventions: Behavioral: Core; Behavioral: App+; Behavioral: App notifications; Behavioral: Buddy
- Experimental Condition #32 (Experimental): core, support calls, app+, buddy, online gym, app notifications
  Interventions: Behavioral: Core; Behavioral: Support Calls; Behavioral: App+; Behavioral: Online gym; Behavioral: App notifications; Behavioral: Buddy

INTERVENTIONS:
Behavioral: Core — The core intervention will include educational materials, access to a basic smartphone app and a Fitbit.
Behavioral: Support Calls — Participants will receive 6 bi-weekly phone calls from study staff.
  Arms: Experimental Condition #1; Experimental Condition #16; Experimental Condition #17; Experimental Condition #18; Experimental Condition #19; Experimental Condition #2; Experimental Condition #20; Experimental Condition #21; Experimental Condition #24; Experimental Condition #27; Experimental Condition #28; Experimental Condition #29; Experimental Condition #3; Experimental Condition #32; Experimental Condition #4; Experimental Condition #5
Behavioral: App+ — Participants will receive "deluxe" version of smartphone app with additional features.
  Arms: Experimental Condition #16; Experimental Condition #17; Experimental Condition #18; Experimental Condition #2; Experimental Condition #22; Experimental Condition #23; Experimental Condition #26; Experimental Condition #27; Experimental Condition #28; Experimental Condition #29; Experimental Condition #31; Experimental Condition #32; Experimental Condition #6; Experimental Condition #7; Experimental Condition #8; Experimental Condition #9
Behavioral: Online gym — Participants will receive access to online exercise videos.
  Arms: Experimental Condition #11; Experimental Condition #13; Experimental Condition #14; Experimental Condition #17; Experimental Condition #19; Experimental Condition #21; Experimental Condition #22; Experimental Condition #23; Experimental Condition #24; Experimental Condition #25; Experimental Condition #26; Experimental Condition #27; Experimental Condition #29; Experimental Condition #32; Experimental Condition #4; Experimental Condition #8
Behavioral: App notifications — Participants will receive motivational app notifications
  Arms: Experimental Condition #12; Experimental Condition #14; Experimental Condition #15; Experimental Condition #18; Experimental Condition #20; Experimental Condition #21; Experimental Condition #23; Experimental Condition #24; Experimental Condition #25; Experimental Condition #26; Experimental Condition #28; Experimental Condition #29; Experimental Condition #31; Experimental Condition #32; Experimental Condition #5; Experimental Condition #9
Behavioral: Buddy — Participants will choose a buddy to receive a Fitbit and support them during the intervention.
  Arms: Experimental Condition #10; Experimental Condition #11; Experimental Condition #12; Experimental Condition #16; Experimental Condition #19; Experimental Condition #20; Experimental Condition #22; Experimental Condition #23; Experimental Condition #24; Experimental Condition #25; Experimental Condition #27; Experimental Condition #28; Experimental Condition #3; Experimental Condition #31; Experimental Condition #32; Experimental Condition #7

SUMMARY:
The overall objective of the proposed research is to pilot test the feasibility and acceptability of a set of more scalable technology-supported physical activity promotion intervention strategies in breast cancer survivors using tMultiphase Optimization Strategy Trial (MOST) methodology. MOST involves highly efficient randomized experimentation to assess the effects of individual intervention strategies, and thereby identify which strategies and what strategy levels make the important contributions to the overall program's effect on physical activity. This information then guides assembly of an optimized physical activity program, that achieves target outcomes with least resource consumption and participant burden. The resulting intervention will have great potential for scalability because it uses technology (smartphones) participants already own and requires no on-site visits.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Stage I-III breast cancer within the last 5 years
2. Have completed last cancer treatment (adjuvant chemotherapy, radiation therapy or surgery) at least 3 months prior to enrollment
3. English speaking
4. Currently participate in less than 60 minutes of moderate and vigorous physical activity per week
5. Own a smartphone
6. Have access to a computer with Internet
7. Participants may be using adjuvant endocrine therapies.
8. Willing to be waitlisted for future wave if current wave reaches capacity

Exclusion Criteria:

-Women will be excluded if they report any of the following:

1. Respiratory, joint or cardiovascular problems precluding physical activity
2. Metastatic disease
3. Planned elective surgery during duration of the intervention/follow-up that would interfere with participation (e.g., breast reconstructive surgery).

ONLY IF PARTICIPATING IN OPTIONAL BLOOD COLLECTION:

1. A prior cardiovascular event (i.e. stroke, myocardial infarction)
2. Have been diagnosed with an acute or chronic immune system medical conditions, or conditions that impact immune and endocrine function (e.g., CFS, Lupus, rheumatoid arthritis, Hepatitis C, or immunosuppressive treatment requiring conditions)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be made available to other researchers in compliance with the NIH Data Sharing Policy.

REFERENCES:
- [Derived] Solk P, Song J, Reading J, Starikovsky J, Cullather E, Wang S, Hasanaj K, Morelli WA, Spring B, Cella D, Penedo F, Ackermann R, Courneya KS, Siddique J, Frey J, Phillips SM. Feasibility and acceptability of the Fit2Thrive mHealth physical activity promotion intervention components in breast cancer survivors. Transl Behav Med. 2025 Jan 16;15(1):ibaf033. doi: 10.1093/tbm/ibaf033. PMID 40795071
- [Derived] Solk P, Song J, Welch WA, Spring B, Cella D, Penedo F, Ackermann R, Courneya KS, Siddique J, Freeman H, Starikovsky J, Mishory A, Alexander J, Wolter M, Carden L, Phillips SM. Effect of the Fit2Thrive Intervention on Patient-reported Outcomes in Breast Cancer Survivors: A Randomized Full Factorial Trial. Ann Behav Med. 2023 Aug 21;57(9):765-776. doi: 10.1093/abm/kaad024. PMID 37203237

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 280 women signed informed consent and enrolled in the study. However, in order to be randomized, participants must complete all baseline assessments. This includes wearing the accelerometer for a minimum of 5 valid days and completing all online questionnaires. A total of 269 women met the criteria for randomization.
Period: Overall Study
Arm/Group | Experimental Condition #1 | Experimental Condition #2 | Experimental Condition #3 | Experimental Condition #4 | Experimental Condition #5 | Experimental Condition #6 | Experimental Condition #7 | Experimental Condition #8 | Experimental Condition #9 | Experimental Condition #10 | Experimental Condition #11 | Experimental Condition #12 | Experimental Condition #13 | Experimental Condition #14 | Experimental Condition #15 | Experimental Condition #16 | Experimental Condition #17 | Experimental Condition #18 | Experimental Condition #19 | Experimental Condition #20 | Experimental Condition #21 | Experimental Condition #22 | Experimental Condition #23 | Experimental Condition #24 | Experimental Condition #25 | Experimental Condition #26 | Experimental Condition #27 | Experimental Condition #28 | Experimental Condition #29 | Experimental Condition #30 | Experimental Condition #31 | Experimental Condition #32
Started | 8 | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 9 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 9 | 8 | 9 | 9 | 8 | 9 | 9 | 8
Completed (Completed the 24 week questionnaires OR had valid data on the accelerometer at 24 weeks) | 7 | 6 | 8 | 8 | 8 | 8 | 9 | 8 | 8 | 7 | 8 | 7 | 7 | 8 | 7 | 8 | 8 | 8 | 7 | 7 | 6 | 7 | 7 | 8 | 8 | 7 | 9 | 7 | 8 | 7 | 8 | 8
Not Completed | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All individuals who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Condition #1 | Experimental Condition #2 | Experimental Condition #3 | Experimental Condition #4 | Experimental Condition #5 | Experimental Condition #6 | Experimental Condition #7 | Experimental Condition #8 | Experimental Condition #9 | Experimental Condition #10 | Experimental Condition #11 | Experimental Condition #12 | Experimental Condition #13 | Experimental Condition #14 | Experimental Condition #15 | Experimental Condition #16 | Experimental Condition #17 | Experimental Condition #18 | Experimental Condition #19 | Experimental Condition #20 | Experimental Condition #21 | Experimental Condition #22 | Experimental Condition #23 | Experimental Condition #24 | Experimental Condition #25 | Experimental Condition #26 | Experimental Condition #27 | Experimental Condition #28 | Experimental Condition #29 | Experimental Condition #30 | Experimental Condition #31 | Experimental Condition #32 | Total
Number analyzed (Participants) | 8 | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 9 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 9 | 8 | 9 | 9 | 8 | 9 | 9 | 8 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (10) | 48.8 (12.2) | 52.4 (9.6) | 58 (5.4) | 54.6 (9.4) | 49 (7.9) | 53.1 (9.8) | 49.1 (7.3) | 50.8 (5.8) | 57.3 (9.9) | 55.6 (12.7) | 52.1 (9.6) | 48.9 (9.1) | 51.3 (9.0) | 53.6 (10.4) | 53.6 (9.1) | 60.4 (9.7) | 54.5 (13.4) | 55.7 (11.3) | 55.1 (7.1) | 54.5 (8.1) | 49.5 (7.2) | 46.9 (13.2) | 60.3 (9.4) | 50.2 (11.3) | 53.1 (8.7) | 53.8 (12.2) | 49.4 (8.6) | 53.1 (13.5) | 52.9 (11) | 50.8 (5.5) | 42.4 (9.1) | 52.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 9 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 9 | 8 | 9 | 9 | 8 | 9 | 9 | 8 | 269
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 19
  Not Hispanic or Latino | 6 | 8 | 8 | 7 | 8 | 9 | 9 | 9 | 9 | 4 | 6 | 7 | 7 | 6 | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 7 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 9 | 9 | 6 | 244
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 16
  White | 5 | 8 | 7 | 6 | 7 | 9 | 9 | 8 | 8 | 4 | 7 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 9 | 7 | 5 | 6 | 7 | 9 | 7 | 7 | 8 | 7 | 9 | 8 | 7 | 234
  More than one race | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 6
Number of Participants Randomized [Count of Participants; unit: Participants] | 8 | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 9 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 9 | 8 | 8 | 9 | 8 | 9 | 8 | 9 | 9 | 8 | 9 | 9 | 8 | 269

OUTCOME MEASURES:

1. Primary Outcome: Adherence to a 12 Week Technology Supported Physical Activity Intervention
Description: Adherence during the 12 week intervention will be monitored continuously using study app. This measures the average percentage of days each participant randomized wore the Fitbit during weeks 1 to 12.
Time Frame: 12 weeks
Population: All participants randomized.
Measure: Mean (Standard Deviation); unit: Percentage of Days Fitbit Worn
Groups:
- All Reporting Groups: All participants randomized regardless of individual randomly assigned combination of On- or Off levels of all intervention factors.
Arm/Group | All Reporting Groups
Number analyzed (Participants) | 269
Percentage of Days Fitbit Worn | 93.0 (12.7)

2. Primary Outcome: Participant Retention
Description: Percentage of participants retained at the end of the 12 week intervention of those randomized [(# of participants randomized who completed at least 1 outcome assessment measure at 12 weeks)/ # randomized*100].
Time Frame: 12 weeks
Measure: Number; unit: Percentage of participants retained
Arm/Group | All Reporting Groups
Number analyzed (Participants) | 269
Percentage of participants retained | 93.3

3. Primary Outcome: Intervention Reach
Description: Percentage of individuals randomized of those who were sent a study screening survey
Time Frame: Baseline
Measure: Number; unit: Percentage of participants randomized
Arm/Group | All Reporting Groups
Number analyzed (Participants) | 269
Percentage of participants randomized | 50.8

4. Secondary Outcome: Change in Moderate to Vigorous Physical Activity From Before to After a 12-Week Intervention
Description: Physical activity will be measured at baseline and at 12 weeks. The ActiGraph accelerometer will be used. At each time point, participants will wear the device for 7 consecutive days during all waking hours, except when bathing or swimming. Each valid minute of wear time will be classified according to intensity (counts/min) using commonly accepted cut-points: sedentary (<100), light activity (100-2019) and moderate/vigorous physical activity (≥2020).
Time Frame: Change from baseline to 12 weeks
Population: One participant was excluded because data values were deemed implausible. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: Minutes per week
Groups:
- Support Calls: Participants receive 6 bi-weekly phone calls from study staff.
- Buddy: Participants choose a buddy to receive a Fitbit and support them during the intervention
- App Notifications: Participants receive motivational app notifications
- Online Gym: Participants receive access to online exercise videos.
- App+: Participants receive "deluxe" version of smartphone app with additional features.
- Core Intervention: Participants receive educational materials, access to a basic smartphone app and a Fitbit.
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core Intervention
Number analyzed (Participants) | 268 | 268 | 268 | 268 | 268 | 268
Minutes per week
  "On" Group Change: number analyzed (Participants) | 133 | 135 | 135 | 132 | 136 | 268
  "On" Group Change | 57.9 (9.4) | 55.5 (9.2) | 59.8 (9.6) | 49.3 (9.0) | 44.3 (8.6) | 53.6 (6.6)
  "Off" Group Change: number analyzed (Participants) | 135 | 133 | 133 | 136 | 132 | 0
  "Off" Group Change | 49.3 (9.0) | 51.7 (9.2) | 47.6 (8.9) | 58.1 (35.0) | 63.5 (9.9) |

5. Secondary Outcome: Change in Moderate to Vigorous Physical Activity From Pre-Intervention to 24-week Follow-up
Description: Physical activity will be measured at baseline and at 24 weeks. The ActiGraph accelerometer will be used. At each time point, participants will wear the device for 7 consecutive days during all waking hours, except when bathing or swimming. Each valid minute of wear time will be classified according to intensity (counts/min) using commonly accepted cut-points: sedentary (<100), light activity (100-2019) and moderate/vigorous physical activity (≥2020).
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Minutes per week
Groups:
- Core: Participants receive educational materials, access to a basic smartphone app and a Fitbit.
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 268 | 268 | 268 | 268 | 268 | 268
Minutes per week
  "On" Group Change: number analyzed (Participants) | 133 | 135 | 135 | 132 | 136 | 268
  "On" Group Change | 28.5 (8.0) | 25.9 (7.9) | 25.3 (7.9) | 15.1 (7.3) | 15.8 (7.4) | 24.6 (5.7)
  "Off" Group Change: number analyzed (Participants) | 135 | 133 | 133 | 136 | 132 | 0
  "Off" Group Change | 49.3 (9.0) | 23.4 (7.8) | 24.0 (7.8) | 58.1 (35.0) | 34.2 (8.4) |

6. Secondary Outcome: Change in Fatigue From Before to After a 12-Week Intervention
Description: Fatigue is measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue 8a health measure. T-scores range from 33.1 to 77.8 Higher scores indicate more fatigue. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Change from baseline to 12 weeks
Population: All participants randomized. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 269 | 269 | 269 | 269 | 269 | 269
t-score on a scale
  "On" Group Change: number analyzed (Participants) | 133 | 135 | 135 | 132 | 137 | 269
  "On" Group Change | -3.1 (0.7) | -3.3 (0.7) | -2.8 (0.7) | -2.2 (0.7) | -2.0 (0.7) | -2.7 (0.5)
  "Off" Group Change: number analyzed (Participants) | 136 | 134 | 134 | 137 | 132 | 0
  "Off" Group Change | -2.3 (0.7) | -2.1 (0.7) | -2.6 (0.7) | -3.2 (0.7) | -3.3 (0.7) |

7. Secondary Outcome: Change in Fatigue From Pre-Intervention to 24-Week Follow-up
Description: Fatigue will be measured at baseline and 24 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue 8a health measure. T-scores range from 33.1 to 77.8 Higher scores indicate more fatigue. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 269 | 269 | 269 | 269 | 269 | 269
t-score on a scale
  "On" Group Change: number analyzed (Participants) | 133 | 135 | 135 | 132 | 137 | 269
  "On" Group Change | -3.5 (0.7) | -4.0 (0.7) | -3.6 (0.7) | -3.3 (0.7) | -3.0 (0.7) | -3.6 (0.5)
  "Off" Group Change: number analyzed (Participants) | 136 | 134 | 134 | 137 | 132 | 0
  "Off" Group Change | -3.7 (0.7) | -3.2 (0.7) | -3.6 (0.7) | -3.9 (0.7) | -4.2 (0.7) |

8. Secondary Outcome: Change in Physical Function From Before to After a 12-Week Intervention
Description: Physical function will be measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-physical function 20a health measure. T-scores range from 32.7 to 62.7. Higher scores indicate better physical functioning. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Change from baseline to 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 269 | 269 | 269 | 269 | 269 | 269
t-score on a scale
  "On" Group Change: number analyzed (Participants) | 133 | 135 | 135 | 132 | 137 | 269
  "On" Group Change | 2.4 (0.4) | 2.3 (0.4) | 2.2 (0.4) | 1.4 (0.4) | 2.5 (0.4) | 2.0 (0.3)
  "Off" Group Change: number analyzed (Participants) | 136 | 134 | 134 | 137 | 132 | 0
  "Off" Group Change | 1.6 (0.4) | 1.7 (0.4) | 1.8 (0.4) | 2.6 (0.4) | 1.5 (0.4) |

9. Secondary Outcome: Treatment Effects for Physical Function From Pre-Intervention to 24-week Follow-up
Description: Physical function will be measured at baseline and 24 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-physical function 20a health measure. T-scores range from 32.7 to 62.7. Higher scores indicate better physical functioning. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population. The treatment effect is calculated as the mean difference in the change in physical function between baseline and 24-weeks for each component on versus off.
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 269 | 269 | 269 | 269 | 269 | 269
t-score on a scale
  "On" Group Change: number analyzed (Participants) | 133 | 135 | 135 | 132 | 137 | 269
  "On" Group Change | 2.2 (0.5) | 2.4 (0.5) | 2.4 (0.5) | 2.0 (0.5) | 2.7 (0.5) | 2.2 (0.3)
  "Off" Group Change: number analyzed (Participants) | 136 | 134 | 134 | 137 | 132 | 0
  "Off" Group Change | 2.0 (0.5) | 2.0 (0.5) | 1.9 (0.4) | 2.4 (0.5) | 1.7 (0.5) |

10. Secondary Outcome: Change in Depression From Before to After a 12-Week Intervention
Description: Depression will be measured at baseline and 12 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-Depression 8a health measure. T-scores range from 38.2 to 81.3. Higher scores indicate more depression. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Change from baseline to 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 269 | 269 | 269 | 269 | 269 | 269
t-score on a scale
  "On" Group Change: number analyzed (Participants) | 133 | 135 | 135 | 132 | 137 | 269
  "On" Group Change | -2.2 (0.6) | -2.2 (0.6) | -2.6 (0.6) | -1.8 (0.6) | -2.1 (0.6) | -2.2 (0.4)
  "Off" Group Change: number analyzed (Participants) | 136 | 134 | 134 | 137 | 132 | 0
  "Off" Group Change | -2.1 (0.6) | -2.1 (0.6) | -1.7 (0.6) | -2.5 (0.6) | -2.2 (0.6) |

11. Secondary Outcome: Change in Depression From Pre-Intervention to 24-week Follow-up
Description: Depression will be measured at baseline and 24 weeks using the Patient Reported Outcomes Measurement Information System (PROMIS)-Depression 8a health measure. T-scores range from 38.2 to 81.3. Higher scores indicate more depression. T-score metric with a mean of 50 and standard deviation of 10 in the U.S. general population.
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Error); unit: t-score on a scale
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 269 | 269 | 269 | 269 | 269 | 269
t-score on a scale
  "On" Group Change: number analyzed (Participants) | 133 | 135 | 135 | 132 | 137 | 269
  "On" Group Change | -1.7 (0.6) | -1.8 (0.6) | -1.6 (0.6) | -1.8 (0.7) | -1.8 (0.6) | -1.8 (0.4)
  "Off" Group Change: number analyzed (Participants) | 136 | 134 | 134 | 137 | 132 | 0
  "Off" Group Change | -1.9 (0.6) | -1.8 (0.6) | -1.9 (0.6) | -1.9 (0.6) | -1.8 (0.6) |

12. Secondary Outcome: Adherence to During the Full 24-Week Study Period
Description: Adherence during the 24-week study period will be monitored continuously using study app. This measure the average percentage of days each randomized participant wore the Fitbit from weeks 1 to 24.
Time Frame: 24 weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Percentage of days the Fitbit was worn
Arm/Group | All Reporting Groups
Number analyzed (Participants) | 269
Percentage of days the Fitbit was worn | 80.0 (25.8)

13. Secondary Outcome: Participant Retention at 24 Week Follow-up
Description: Percentage of participants retained at 24 weeks of those randomized
Time Frame: 24 weeks
Population: All participants randomized
Measure: Number; unit: Percentage of participants retained
Arm/Group | All Reporting Groups
Number analyzed (Participants) | 269
Percentage of participants retained | 90

14. Secondary Outcome: Change in Interleukin-6 (IL-6) From Before to After a12 Week Intervention (Optional)
Description: Interleukin-6 (IL-6) will be self-collected via finger prick to obtain dried blood spot and will be quantified using a standard multiplex electrochemiluminescent immunoassay protocol.
Time Frame: Change from baseline to 12 weeks
Population: This includes all participants who agreed to participate in dried blood spots and had at least one valid sample for IL-6. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 121 | 121 | 121 | 121 | 121 | 121
pg/mL
  "On" Group Change: number analyzed (Participants) | 52 | 62 | 59 | 57 | 57 | 121
  "On" Group Change | -0.07 (0.10) | -0.06 (0.09) | -0.05 (0.09) | -0.08 (0.10) | 0.01 (0.09) | -0.02 (0.06)
  "Off" Group Change: number analyzed (Participants) | 69 | 59 | 62 | 64 | 64 | 0
  "Off" Group Change | 0.02 (0.08) | 0.02 (0.09) | 0.01 (0.09) | 0.05 (0.07) | -0.06 (0.09) |

15. Secondary Outcome: Change in Interleukin-6 (IL-6) From Pre-Intervention to 24-week Follow-up (Optional)
Description: Interleukin-6 (IL-6) will be self-collected via finger prick to obtain dried blood spot and will be quantified using a standard multiplex electrochemiluminscent immunoassay protocol.
Time Frame: Change from baseline to 24 weeks
Population: This includes all participants who agreed to participate in dried blood spots and had at least one valid sample for IL-6.In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 121 | 121 | 121 | 121 | 121 | 121
pg/mL
  "On" Group Change: number analyzed (Participants) | 52 | 62 | 59 | 57 | 57 | 121
  "On" Group Change | 0.14 (0.10) | 0.13 (0.10) | 0.09 (0.10) | 0.06 (0.11) | 0.17 (0.10) | 0.14 (0.07)
  "Off" Group Change: number analyzed (Participants) | 69 | 59 | 62 | 64 | 64 | 0
  "Off" Group Change | 0.14 (0.09) | 0.15 (0.09) | 0.18 (0.09) | 0.22 (0.08) | 0.10 (0.09) |

16. Secondary Outcome: Change in Interleukin-10 (IL-10) From Before to After a 12 Week Intervention (Optional)
Description: Interleukin-10 (IL-10) will be self-collected via finger prick to obtain dried blood spot and will be quantified using a standard multiplex electrochemiluminscent immunoassay protocol.
Time Frame: Change from baseline to 12 weeks
Population: This includes all participants who agreed to participate in dried blood spots and had at least one valid sample for IL-10. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 121 | 121 | 121 | 121 | 121 | 121
pg/mL
  "On" Group Change: number analyzed (Participants) | 52 | 62 | 59 | 57 | 57 | 121
  "On" Group Change | 0.03 (0.03) | -0.01 (0.03) | -0.01 (0.03) | -0.02 (0.04) | 0.03 (0.03) | 0 (0.02)
  "Off" Group Change: number analyzed (Participants) | 69 | 59 | 62 | 64 | 64 | 0
  "Off" Group Change | 0.12 (0.05) | 0.01 (0.03) | 0 (0.03) | 0.02 (0.03) | -0.03 (0.03) |

17. Secondary Outcome: Change in Interleukin-10 (IL-10) From Pre-Intervention to 24-week Follow-up (Optional)
Description: Interleukin-10 (IL-10) will be self-collected via finger prick to obtain dried blood spot and will be quantified using a standard multiplex electrochemiluminscent immunoassay protocol. Higher IL-10 may have protective effects.
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 121 | 121 | 121 | 121 | 121 | 121
pg/mL
  "On" Group Change: number analyzed (Participants) | 52 | 62 | 59 | 57 | 57 | 121
  "On" Group Change | 0.11 (0.04) | 0.04 (0.03) | 0.06 (0.04) | 0.06 (0.04) | 0.08 (0.04) | 0.05 (0.02)
  "Off" Group Change: number analyzed (Participants) | 69 | 59 | 62 | 64 | 64 | 0
  "Off" Group Change | -0.01 (0.03) | 0.07 (0.03) | 0.05 (0.04) | 0.04 (0.03) | 0.02 (0.03) |

18. Secondary Outcome: Change in Tumor Necrosis Factor-alpha (TNFα) From Before to After a12 Week Intervention (Optional)
Description: tumor necrosis factor-alpha (TNFα) will be self-collected via finger prick to obtain dried blood spot and will be quantified using a standard multiplex electrochemiluminscent immunoassay protocol. Lower values are better.
Time Frame: Change from baseline to 12 weeks
Population: This includes all participants who agreed to participate in dried blood spots and had at least one valid sample for TNFα. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 121 | 121 | 121 | 121 | 121 | 121
pg/mL
  "On" Group Change: number analyzed (Participants) | 52 | 62 | 59 | 57 | 57 | 121
  "On" Group Change | 0.22 (0.17) | -0.27 (0.15) | -0.11 (0.16) | -0.27 (0.17) | -0.17 (0.17) | -0.13 (0.11)
  "Off" Group Change: number analyzed (Participants) | 69 | 59 | 62 | 64 | 64 | 0
  "Off" Group Change | -0.05 (0.14) | 0.01 (0.15) | -0.15 (0.15) | 0.01 (0.13) | -0.10 (0.15) |

19. Secondary Outcome: Change in Tumor Necrosis Factor-alpha (TNFα) From Pre-Intervention to 24-week Follow-up (Optional)
Description: tumor necrosis factor-alpha (TNFα) will be self-collected via finger prick to obtain dried blood spot and will be quantified using a standard multiplex electrochemiluminscent immunoassay protocol. TLower values are better.
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 18
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 121 | 121 | 121 | 121 | 121 | 121
pg/mL
  "On" Group Change: number analyzed (Participants) | 52 | 62 | 59 | 57 | 57 | 121
  "On" Group Change | 0.22 (0.17) | 0.14 (0.16) | 0.07 (0.17) | -0.03 (0.18) | 0.24 (0.17) | 0.09 (0.11)
  "Off" Group Change: number analyzed (Participants) | 69 | 59 | 62 | 64 | 64 | 0
  "Off" Group Change | -0.05 (0.14) | 0.03 (0.15) | 0.11 (0.15) | 0.20 (0.13) | -0.07 (0.14) |

20. Secondary Outcome: Change in C-reactive Protein (CRP) From Before to After a12 Week Intervention (Optional)
Description: C-reactive protein (CRP) will be self-collected via finger prick to obtain dried blood spot and will be quantified using ELISA. Lower values are better.
Time Frame: Change from baseline to 12 weeks
Population: This includes all participants who agreed to participate in dried blood spots and had at least one valid sample for CRP. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 199 | 199 | 199 | 199 | 199 | 199
mg/L
  "On" Group Change: number analyzed (Participants) | 94 | 103 | 104 | 96 | 97 | 199
  "On" Group Change | -0.04 (0.19) | -0.14 (0.18) | 0.14 (0.18) | 0.22 (0.19) | -0.02 (0.19) | 0.07 (0.13)
  "Off" Group Change: number analyzed (Participants) | 105 | 96 | 95 | 103 | 102 | 0
  "Off" Group Change | 0.18 (0.18) | 0.28 (0.19) | 0 (0.19) | -0.08 (0.18) | 0.16 (0.18) |

21. Secondary Outcome: Change in C-reactive Protein (CRP) From Pre-Intervention to 24-week Follow-up (Optional)
Description: C-reactive protein (CRP) will be self-collected via finger prick to obtain dried blood spot and will be quantified using standard ELISA. Lower values are better.
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 20
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 199 | 199 | 199 | 199 | 199 | 199
mg/L
  "On" Group Change: number analyzed (Participants) | 94 | 103 | 104 | 96 | 97 | 199
  "On" Group Change | 0.05 (0.20) | -0.09 (0.18) | -0.06 (0.18) | 0.01 (0.26) | -0.07 (0.19) | -0.09 (0.13)
  "Off" Group Change: number analyzed (Participants) | 105 | 96 | 95 | 103 | 102 | 0
  "Off" Group Change | -0.22 (0.18) | -0.09 (0.19) | -0.12 (0.19) | -0.21 (0.18) | -0.10 (0.18) |

22. Secondary Outcome: Change in Triglycerides From Before to After a 12 Week Intervention (Optional)
Description: Triglycerides are self-collected via finger prick to obtain a dried blood spot and quantified using a standard coupled enzymatic protocol.
Time Frame: Change from baseline to 12 weeks
Population: This includes all participants who agreed to participate in dried blood spots and had at least one valid sample for triglycerides. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 146 | 146 | 146 | 146 | 146 | 146
mg/dL
  "On" Group Change: number analyzed (Participants) | 66 | 80 | 69 | 70 | 73 | 146
  "On" Group Change | -17.35 (23.23) | 6.63 (20.99) | -14.96 (22.55) | 28.08 (22.52) | 9.01 (21.33) | 4.40 (15.28)
  "Off" Group Change: number analyzed (Participants) | 80 | 66 | 77 | 76 | 73 | 0
  "Off" Group Change | 25.43 (19.72) | 1.45 (21.97) | 23.04 (20.63) | -20.00 (20.42) | -0.93 (21.46) |

23. Secondary Outcome: Change in Triglycerides From Pre-Intervention to 24-week Follow-up (Optional)
Description: Triglycerides are self-collected via finger prick to obtain a dried blood spot and quantified using a standard coupled enzymatic protocol. Lower values are better.
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 22
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 146 | 146 | 146 | 146 | 146 | 146
mg/dL
  "On" Group Change: number analyzed (Participants) | 66 | 80 | 69 | 70 | 73 | 146
  "On" Group Change | -10.81 (23.82) | 5.15 (21.59) | 3.60 (24.16) | 17.12 (23.82) | 20.99 (22.32) | 16.10 (15.80)
  "Off" Group Change: number analyzed (Participants) | 80 | 66 | 77 | 76 | 73 | 0
  "Off" Group Change | 43.01 (20.76) | 27.05 (22.82) | 28.60 (20.68) | 15.09 (20.69) | 11.21 (22.00) |

24. Secondary Outcome: Change in Blood Glucose From Before to After a 12 Week Intervention (Optional)
Description: Blood glucose is self-collected via finger prick to obtain a dried blood spot and quantified using a standard coupled enzymatic protocol.
Time Frame: Change from baseline to 12 weeks
Population: This includes all participants who agreed to participate in dried blood spots and had at least one valid sample for blood glucose. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 162 | 162 | 162 | 162 | 162 | 162
mg/dL
  "On" Group Change: number analyzed (Participants) | 73 | 89 | 84 | 76 | 78 | 162
  "On" Group Change | 1.16 (3.2) | 3.90 (2.99) | 2.68 (3.07) | 3.83 (3.20) | 3.29 (3.16) | 2.62 (2.11)
  "Off" Group Change: number analyzed (Participants) | 89 | 73 | 78 | 86 | 84 | 0
  "Off" Group Change | 4.06 (2.76) | 1.34 (3.05) | 2.56 (2.93) | 1.40 (2.79) | 1.94 (2.84) |

25. Secondary Outcome: Change in Blood Glucose From Pre-Intervention to 24-week Follow-up (Optional)
Description: as for outcome 24
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 162 | 162 | 162 | 162 | 162 | 162
mg/dL
  "On" Group Change: number analyzed (Participants) | 73 | 89 | 84 | 76 | 78 | 162
  "On" Group Change | -3.13 (3.45) | -3.03 (3.19) | -1.33 (3.43) | -1.20 (3.53) | 0.38 (3.38) | -1.55 (2.31)
  "Off" Group Change: number analyzed (Participants) | 89 | 73 | 78 | 86 | 84 | 0
  "Off" Group Change | 0.04 (3.03) | -0.06 (3.30) | -1.76 (3.06) | -1.89 (2.96) | -3.47 (3.11) |

26. Secondary Outcome: Change in High Density Lipoprotein Cholesterol (HDL) From Before to After a12 Week Intervention (Optional)
Description: High density lipoprotein cholesterol (HDL) is self-collected via finger prick to obtain a dried blood spot and quantified using a standard coupled enzymatic protocol.
Time Frame: Change from baseline to 12 weeks
Population: This includes all participants who agreed to participate in dried blood spots and had at least one valid sample for HDL. In a full factorial trial, participants are randomized to receive each intervention component (support calls, buddy, app notifications, online gym, app+) "on" or "off." Participants randomized to "on" are compared to those randomized to "off." All participants get the core intervention so there is no comparison group.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 177 | 177 | 177 | 177 | 177 | 177
mg/dL
  "On" Group Change: number analyzed (Participants) | 78 | 95 | 88 | 84 | 87 | 177
  "On" Group Change | 0.37 (4.20) | 3.43 (3.87) | 5.19 (3.98) | 1.18 (4.11) | 3.91 (4.05) | 0.31 (2.78)
  "Off" Group Change: number analyzed (Participants) | 99 | 82 | 89 | 93 | 90 | 0
  "Off" Group Change | -1.00 (3.67) | -4.05 (4.00) | -5.82 (3.87) | 0.55 (3.74) | -4.53 (3.83) |

27. Secondary Outcome: Change in High Density Lipoprotein Cholesterol (HDL) From Pre-Intervention to 24-week Follow-up(Optional)
Description: as for outcome 26
Time Frame: Change from baseline to 24 weeks
Population: as for outcome 26
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Support Calls | Buddy | App Notifications | Online Gym | App+ | Core
Number analyzed (Participants) | 177 | 177 | 177 | 177 | 177 | 177
mg/dL
  "On" Group Change: number analyzed (Participants) | 78 | 95 | 88 | 84 | 87 | 177
  "On" Group Change | 2.72 (4.25) | 0.59 (3.91) | 2.01 (4.27) | 0.51 (4.37) | 4.50 (4.28) | 0.57 (2.91)
  "Off" Group Change: number analyzed (Participants) | 99 | 82 | 89 | 93 | 90 | 0
  "Off" Group Change | -1.58 (3.94) | 0.55 (4.29) | -0.86 (3.93) | 0.64 (3.83) | -3.36 (3.92) |

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the 24 week study period.
Arm/Group | Experimental Condition #1 | Experimental Condition #2 | Experimental Condition #3 | Experimental Condition #4 | Experimental Condition #5 | Experimental Condition #6 | Experimental Condition #7 | Experimental Condition #8 | Experimental Condition #9 | Experimental Condition #10 | Experimental Condition #11 | Experimental Condition #12 | Experimental Condition #13 | Experimental Condition #14 | Experimental Condition #15 | Experimental Condition #16 | Experimental Condition #17 | Experimental Condition #18 | Experimental Condition #19 | Experimental Condition #20 | Experimental Condition #21 | Experimental Condition #22 | Experimental Condition #23 | Experimental Condition #24 | Experimental Condition #25 | Experimental Condition #26 | Experimental Condition #27 | Experimental Condition #28 | Experimental Condition #29 | Experimental Condition #30 | Experimental Condition #31 | Experimental Condition #32
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/8 | 0/9 | 1/9 | 0/9 | 0/9 | 0/9 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/9 | 0/8 | 0/8 | 0/9 | 0/8 | 0/9 | 1/8 | 0/9 | 0/9 | 0/8 | 0/9 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/8 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/9 | 0/8 | 0/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9 | 0/9 | 0/8 | 0/9 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 3/9 | 1/8 | 1/8 | 0/9 | 1/9 | 1/9 | 0/9 | 2/9 | 0/8 | 1/8 | 1/8 | 0/8 | 1/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 2/9 | 0/8 | 0/8 | 0/9 | 2/8 | 0/9 | 1/8 | 1/9 | 2/9 | 0/8 | 0/9 | 1/9 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Condition #1 (N=8) | Experimental Condition #2 (N=9) | Experimental Condition #3 (N=8) | Experimental Condition #4 (N=8) | Experimental Condition #5 (N=9) | Experimental Condition #6 (N=9) | Experimental Condition #7 (N=9) | Experimental Condition #8 (N=9) | Experimental Condition #9 (N=9) | Experimental Condition #10 (N=8) | Experimental Condition #11 (N=8) | Experimental Condition #12 (N=8) | Experimental Condition #13 (N=8) | Experimental Condition #14 (N=8) | Experimental Condition #15 (N=8) | Experimental Condition #16 (N=8) | Experimental Condition #17 (N=8) | Experimental Condition #18 (N=8) | Experimental Condition #19 (N=8) | Experimental Condition #20 (N=9) | Experimental Condition #21 (N=8) | Experimental Condition #22 (N=8) | Experimental Condition #23 (N=9) | Experimental Condition #24 (N=8) | Experimental Condition #25 (N=9) | Experimental Condition #26 (N=8) | Experimental Condition #27 (N=9) | Experimental Condition #28 (N=9) | Experimental Condition #29 (N=8) | Experimental Condition #30 (N=9) | Experimental Condition #31 (N=9) | Experimental Condition #32 (N=8)
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Torn/Pulled Muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendinitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple Sclerosis Relapse (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast reconstruction surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness Spell (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Concussion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sprain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03131440/Prot_SAP_000.pdf